CLINICAL TRIAL: NCT01176422
Title: Telomere and Telomerase
Status: Withdrawn | Type: Observational
Why Stopped: lack of resources; no patient enrollment
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12016
Record Dates: First submitted 2010-08-03; First posted 2010-08-06 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Two teaspoons of blood will be collected - one teaspoon before subject begins treatment for disease and one teaspoon will be collected when subject completes treatment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- advanced Myelodysplastic Syndrome or acute myeloid leukemia: advanced MDS and AML with/without associated cytogenetic abnormality
  Interventions: Genetic: Blood sample

INTERVENTIONS:
Genetic: Blood sample — Blood samples will be collected before and after treatment completion.

SUMMARY:
Researchers hope to determine if the DNA is shortened in your body and determine if there is an increase in the protein that shortens DNA called telomerase.

DETAILED DESCRIPTION:
A telomere is a region of repetitive DNA at the end of chromosomes, which protects the end of the chromosome from destruction. Telomeres can be viewed as the tips on the ends of shoelaces that keep them from unraveling. Telomeres compensate for incomplete semi-conservative DNA replication at chromosomal ends. In absence of a reparative process, DNA sequences would be lost in every replicative phase until they reached a critical level, at which point cell division would stop.

Loss of telomeres leads to chromosome end-to-end fusion, chromosome re-arrangements, and genome instability.

Telomerase is a "ribonucleoprotein complex" composed of a protein component and an RNA primer sequence which acts to protect the terminal ends of chromosomes. Telomerase is the natural enzyme which promotes telomere repair. It is however not active in most cells. It certainly is active though in stem cells, germ cells, hair follicles and in 90 percent of cancer cells. Telomerase functions by adding bases to the ends of the telomeres. As a result of this telomerase activity, these cells seem to possess a kind of immortality.

Progressive shortening or attrition of telomere length with consequent genomic instability leading to cancer has been described in various hematological malignancies including acute and chronic myeloid leukemia.

Reduced telomere length has been documented in patients with the progressive BM failure syndrome called Dyskeratosis Congenita. Abnormalities in these patients include skin pigmentation, nail dystrophy and leukoplakia. Mutations in the telomere maintenance mechanism have been implicated in the pathogenesis of this heterogeneous condition.

Myelodysplastic syndrome is an acquired clonal stem cell disorder characterized by in-effective hematopoiesis, increased intra-medullary apoptosis and peripheral cytopenia. A number of such patients will eventually develop worsening cytopenia evolving into acute myeloid leukemia. A number of studies have investigated telomerase activity and telomere length in patients with MDS and AML. Telomere shortening was significantly more pronounced in patients with cytogenetic alterations as compared to patients with normal karyotypes.

Genomic instability develops with progressive telomere shortening. The Telomere attrition related genome instability is a stress that leads to up-regulation of specified DNA damage foci. These telomere-associated DNA damage points are often called as Telomere Dysfunction-Induced Focus (TIF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Myelodysplastic Syndrome (MDS) or acute myeloid leukemia
* must be 18 years of age
* must be able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the BMT/Hematology clinic in the Cancer Center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Identification and resolution of telomere dysfunction-induced focus (TIF) and normalization of telomerase activity | up to 24 weeks
  Advancing myelodysplasia is associated with progressive telomere attrition and clonal chromosomal evolution. Based on this hypothesis, we expect to see identification of TIF by immunostaining and increase in Telomerase activity in peripheral blood granulocytes of patients with advanced Myelodysplastic Syndrome (MDS) and acute myeloid leukemia.
  We also expect to see resolution of TIF and normalization of telomerase activity upon treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Ganguly, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Westwood Campus, Westwood, Kansas, United States